CLINICAL TRIAL: NCT02305342
Title: Antibiotic Susceptibility of Bacterial Uro-Pathogens In Patients Attending Family Physicians" (In Vitro Study)
Brief Title: Sensitivity of Antibiotics for Urinary Tract Infections Patients Attending Family Physicians
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: ENOX5001
Record Dates: First submitted 2014-11-17; First posted 2014-12-02 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Urinary Tract Infections (UTIs)
Keywords: Uncomplicated UTI; Enoxacin
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Urinary Tract Infections (UTIs): Uncomplicated UTIs

SUMMARY:
This study is aiming to evaluate the sensitivity of uropathogens isolated in patients with community acquired UTI with Enoxacin in comparison to other antimicrobials. While Secondary objective is to study the spectrum of uropathogens responsible for community acquired UTI in local population

DETAILED DESCRIPTION:
Mid stream , clean catch urine specimens of patients with uncomplicated community acquired UTI sent to microbiology labs by treating consultants from filter clinics for evaluation of pathogens will be utilized for sensitivity analysis.

Only the first positive urine culture obtained per sample will be included in the analysis to eliminate any possibility of recurrence and nosocomial infection. The polymicrobial cultures and cultures with multidrug-resistant uropathogens will not be included in the analysis. Cultures with common contaminants, including coagulase-negative staphylococci and hemolytic streptococci, and cultures with Candida growth will be excluded. .

Data points to be collected will be date of collection, computer generated Lab #, age, gender,list of cultured organisms, sensitivity of organisms with antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Samples from primary care clinics from patients who reports UTI symptoms and in which uropathogens are isolated will be included.

Exclusion Criteria:

* Samples from specialized, hospitalized or catheterized patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinics
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Uropathogens | 3 months
  Sensitivity of identified organisms shall be noted by the zone size in millimeters of the cultured organisms. "Sensitive", "Intermediate" and "Resistant" labels shall be used as per Clinical Laboratory Standard Institute (CLSI) guidelines.

SECONDARY OUTCOMES:
Common UTI pathogens | 3 months
  To enlist the number and names of identified uropathogens from urine cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Raeefuddin Ahmed, MBBS, FCPS, Study Director — Abbott
Locations (1):
- Research facility ID ORG-001126, Karachi, Pakistan